CLINICAL TRIAL: NCT07287722
Title: Clinical and Biochemical Assessment of the Soft Tissue Response to Printed Versus Milled Polymethyl Methacrylate Custom Healing Abutments
Brief Title: Soft Tissue Response and IL-1β Levels Around CAD/CAM-Milled vs 3D-Printed PMMA Healing Abutments
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Hassan Eid Toto (Other)
Responsible Party: Sponsor-Investigator, Ali Hassan Eid Toto, MSC Candidate in periodontology department Alexandria university, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AlexandriaUali
Record Dates: First submitted 2025-11-23; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Peri-implant Soft Tissue Healing
Keywords: Dental implants; Healing abutments; PMMA; CAD/CAM milled abutments; 3D-printed abutments; Peri-implant soft tissue; Peri-implant inflammation; Interleukin-1 beta (IL-1β); Peri-implant crevicular fluid; Surface roughness; Degree of conversion; Biocompatibility; Digital dentistry; Soft tissue healing

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to one of two parallel groups. Each participant receives only one type of healing abutment either a CAD/CAM-milled PMMA abutment or a 3D-printed PMMA abutment at the time of second-stage implant surgery and remains in that assigned group throughout the 4-week follow-up period. No crossover occurs between groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM-Milled PMMA Healing Abutment (Experimental): Participants receive a customized PMMA healing abutment manufactured using CAD/CAM milling from a pre-polymerized PMMA block. The abutment is attached to the implant at second-stage surgery to guide soft-tissue healing.
  Interventions: Device: CAD/CAM-Milled PMMA Healing Abutment
- 3D-Printed PMMA Healing Abutment (Experimental): Participants receive a customized PMMA healing abutment manufactured using 3D printing from a light-cured PMMA resin, followed by post-processing and UV curing. The abutment is attached to the implant at second-stage surgery.
  Interventions: Device: 3D-Printed PMMA Healing Abutment

INTERVENTIONS:
Device: CAD/CAM-Milled PMMA Healing Abutment — A customized healing abutment fabricated by subtractive CAD/CAM milling from a pre-polymerized PMMA block. Milling produces a highly polished, low-porosity surface with a high degree of polymerization. The abutment is connected to a Ti-base and placed at second-stage surgery to shape peri-implant soft tissues.
  Arms: CAD/CAM-Milled PMMA Healing Abutment
Device: 3D-Printed PMMA Healing Abutment — A customized healing abutment produced by additive manufacturing (3D printing) using a light-cured PMMA resin. The abutment is printed layer-by-layer, washed in isopropyl alcohol, UV-cured, finished, and polished. This manufacturing technique results in a different surface texture and polymerization level compared to milled PMMA. The abutment is attached to a Ti-base and placed at second-stage surgery.
  Arms: 3D-Printed PMMA Healing Abutment

SUMMARY:
This study looked at how the gums and tissues around dental implants heal when using two different types of temporary healing caps made of PMMA (a common dental material). These healing caps help shape the gums before placing the final crown.

There are two ways to make these caps:

1. CAD/CAM-milled (carved from a solid block)
2. 3D-printed (built layer by layer using resin) The goal was to find out which type leads to healthier gum tissue. What the Researchers Did

   * 22 dental implants in 22 patients were included.
   * Each implant received one healing cap-either milled or 3D-printed.
   * Patients were checked after 1 week, 2 weeks, and 4 weeks.
   * The team measured:

     * Gum inflammation
     * Bleeding around the implant
     * Plaque buildup
     * Pocket depth around the implant
     * Levels of an inflammatory marker called Interleukin-1β (IL-1β) in the gum fluid (higher levels mean more inflammation).
     * Surface smoothness and material quality of each type of healing cap. What the Study Found
   * Gum inflammation and bleeding were higher with 3D-printed caps, especially at week 4.
   * IL-1β levels were much higher around 3D-printed caps-showing more inflammation.
   * Both types had some increase in plaque and probing depth over time, but there was no major difference between groups.
   * The milled caps had smoother surfaces and better material quality, which may have helped reduce irritation and inflammation.
   * 3D-printed caps were rougher and had lower polymerization (more leftover monomers), which may trigger soft-tissue irritation.

What This Means

* CAD/CAM-milled PMMA healing caps appear to be safer and healthier for gum healing around dental implants.
* They may help reduce early inflammation, support better tissue health, and more predictably shape the gums during healing.

Why This Matters for Patients

* Using a smoother, better-finished healing cap may lower the risk of early gum inflammation.
* Healthier soft tissue around an implant leads to better long-term implant stability.
* This information can help dentists choose the best healing cap for optimal healing.

Study Timeframe

• The follow-up was 4 weeks, so results focus on early healing. More research is needed to know long-term differences.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25 to 65 years
* Presence of one osseointegrated dental implant placed at least 8 weeks prior to second-stage surgery
* Adequate zone of attached keratinized gingiva (> 1 mm) around the implant site
* Good general health and able to provide informed consent
* Willing and able to attend all follow-up visits (1, 2, and 4 weeks)

Exclusion Criteria:

* Smoking more than 20 cigarettes per day
* Presence of systemic diseases that may affect healing (e.g., autoimmune conditions, uncontrolled diabetes, immunosuppressive disorders)
* Oral inflammatory conditions or active oral infections
* History of head and neck radiation therapy or chemotherapy
* Use of corticosteroids or antibiotics within the last 3 months
* Parafunctional habits (e.g., bruxism)
* Pregnant or breastfeeding individuals
* Implants with insufficient attached gingiva or poor oral hygiene maintenance

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2025-11-23 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Interleukin-1β (IL-1β) Level in Peri-Implant Crevicular Fluid | up to 4 weeks
  Concentration of IL-1β in peri-implant crevicular fluid collected using sterile paper points. Samples are stored at -80°C and analyzed using ELISA kits. Higher IL-1β levels indicate greater inflammatory response. Mean IL-1β values are compared between CAD/CAM-milled and 3D-printed PMMA healing abutment groups at each time point.

SECONDARY OUTCOMES:
Modified Gingival Index (MGI) | up to 4 weeks
  Soft-tissue inflammation around the healing abutment assessed using the Modified Gingival Index (0-3 scale) at four peri-implant sites (mesial, distal, buccal, palatal). Higher scores indicate more severe inflammation. Group differences and changes over time are evaluated.
Plaque Index (PI) | up to 4 weeks
  Plaque accumulation measured at four implant surfaces using a 0-3 scale (0 = no plaque; 3 = heavy soft deposits). Mean PI values are compared between study groups and across time points.
Bleeding on Probing (BOP) | up to 4 weeks
  Presence or absence of bleeding upon gentle probing around the healing abutment. BOP is recorded as a binary variable and expressed as the percentage of implants with bleeding in each group.
Probing Pocket Depth (PPD) | up to 4 weeks
  Probing depth in millimeters measured at four peri-implant sites using a plastic periodontal probe. Mean pocket depths and changes over time are compared between groups.
Surface Roughness of PMMA Healing Abutments | Immediately after fabrication
  Surface roughness parameters (Ra, Rz, Rp, Rv) measured via profilometry for CAD/CAM-milled and 3D-printed PMMA abutments. Higher values indicate rougher surfaces. Group means are compared.
Degree of Conversion (%) of PMMA Material | Immediately after fabrication
  Degree of polymerization of PMMA material measured using spectroscopic methods. Higher percentages indicate more complete polymerization and lower residual monomer content. Compared between milled and 3D-printed groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No